CLINICAL TRIAL: NCT04643158
Title: A Two-part Phase IIa Randomised, Double-blind, Placebo-controlled, Dose-ranging, Multi-centre Study to Assess Efficacy and Safety of Inhaled AZD1402 Administered as a Dry Powder for Four Weeks in Adults With Asthma on Medium-to-High Dose Inhaled Corticosteroids
Brief Title: Efficacy and Safety of Inhaled AZD1402 Administered for Four Weeks in Adults With Asthma on Medium-to-High Dose Inhaled Corticosteroids
Acronym: APATURA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The decision was based on lung findings from a non-clinical 13-week Good Laboratory Practice (GLP) toxicology study, which are not a concern for the active clinical studies but do not support long-term use and progression to later-stage development.
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D2912C00003; 2020-002828-37 (EudraCT Number)
Record Dates: First submitted 2020-11-23; First posted 2020-11-24 (Actual); Results first posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Asthma
Keywords: AZD1402; placebo; Anticalin® protein; dry powder inhaler; inhaled corticosteroids; efficacy; safety
MeSH Terms: conditions — Asthma | interventions — 3-(2-(4-azidobenzamidino)ethyl)-5-hydroxyindole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part 1 and Part 2: AZD1402 Dose 1 (Experimental): Randomised participants will receive oral inhalation of AZD1402 Dose 1 via DPI.
  Interventions: Drug: AZD1402; Drug: Short acting beta agonist (SABA) (rescue medication); Drug: Run-in medications (ICS-LABA combination)
- Part 1 and Part 2: AZD1402 Dose 2 (Experimental): Randomised participants will receive oral inhalation of AZD1402 Dose 2 via DPI.
  Interventions: Drug: AZD1402; Drug: Short acting beta agonist (SABA) (rescue medication); Drug: Run-in medications (ICS-LABA combination)
- Part 1: AZD1402 Dose 3 (Experimental): Randomised participants will receive oral inhalation of AZD1402 Dose 3 via DPI.
  Interventions: Drug: AZD1402; Drug: Short acting beta agonist (SABA) (rescue medication); Drug: Run-in medications (ICS-LABA combination)
- Part 1 and Part 2: Placebo (Placebo Comparator): Randomised participants will receive oral inhalation of matching placebo via DPI.
  Interventions: Drug: Placebo; Drug: Short acting beta agonist (SABA) (rescue medication); Drug: Run-in medications (ICS-LABA combination)

INTERVENTIONS:
Drug: AZD1402 — Randomised participants will receive oral inhalation of AZD1402, via DPI.
  Arms: Part 1 and Part 2: AZD1402 Dose 1; Part 1 and Part 2: AZD1402 Dose 2; Part 1: AZD1402 Dose 3
Drug: Placebo — Randomised participants will receive oral inhalation of matching placebo via DPI.
  Arms: Part 1 and Part 2: Placebo
Drug: Short acting beta agonist (SABA) (rescue medication) — In addition to study intervention, all participants will be provided with a SABA as rescue medication (eg, salbutamol/albuterol), to be used throughout the Run-in and Treatment Periods. All participants should refrain from taking a SABA as rescue medication 6 hours prior to pulmonary function tests.
  Dosage levels: 100 μg per nominal dose 90 μg per nominal dose pro re nata (as required) (PRN)
Drug: Run-in medications (ICS-LABA combination) — During the Run-in Period, the participants are required to maintain on their ICS-LABA dose. Controller medications (eg, ICS LABA) should remain at a stable dose and be taken after study intervention as applicable.
  These drugs are used as standard of care.

SUMMARY:
This is a randomised, placebo-controlled, double-blinded, multi-centre, 2-part study to assess the efficacy and safety of inhaled AZD1402. Part 1 will be performed in a Lead-in Cohort for each dose level to evaluate the safety and pharmacokinetics (PK) in a population with asthma controlled on medium dose inhaled corticosteroids (ICS)-long acting beta agonists (LABA) before progressing to dosing in adults with asthma who are uncontrolled on medium-to-high dose ICS-LABA in Part 2. The study will recruit participants receiving treatment with medium dose ICS with LABA for Part 1 and participants receiving treatment with medium-to-high dose ICS with LABA for Part 2 (separate inhalers or combination product).

Part 2 will be initiated following evaluation of safety and PK at the relevant dose level in Part 1a. The entire study period for each participant in both Parts 1 and 2, is approximately 3.5 months; a 2-week Screening Period, a 4 week Run-in Period, 4 weeks of Treatment Period, and 4 weeks of Follow-Up Period.

DETAILED DESCRIPTION:
Part 1 of the study will be randomised, double blind, placebo-controlled, and conducted in parallel for the 2 lower dose levels (Part 1a) followed by an unblinded safety review and escalation to the highest dose (Part 1b) dependent on the outcome of the safety review.

Part 1a will consist of 30 participants who will be randomised 1:1:1 to receive 1 of the 2 lower AZD1402 dry power inhaler (DPI) doses (Dose 1 or Dose 2) or placebo in parallel. Part 1b will consist of 15 participants who will be randomised 2:1 to receive the highest AZD1402 DPI dose (Dose 3) or placebo.

Part 1a Lead-in Cohort

* AZD1402 Dose 1
* AZD1402 Dose 2
* Placebo

Part 1b Lead-in Cohort

* AZD1402 Dose 3
* Placebo

Part 2 will be randomised, double blind, placebo controlled and will include approximately 165 participants randomised 2:1 (active to placebo) to evaluate 2 inhaled dose levels of AZD1402 versus placebo.

Part 2 will be started after the unblinded safety review for Part 1a. Part 2 will include:

* AZD1402 Dose 1
* AZD1402 Dose 2
* Placebo

ELIGIBILITY:
Inclusion Criteria:

* Participants who have a documented clinical diagnosis of asthma for ≥ 12 months before Visit 1.
* Participants who are able to perform acceptable pulmonary function testing for FEV1.
* Participants who are able to demonstrate the ability to use the study inhalation device properly.
* Male participants must be surgically sterile or agree to use highly-effective contraceptives.
* All female participants must have a negative serum pregnancy test at Screening. Female participants of non-childbearing potential, Female participants of childbearing potential must have a negative urine pregnancy test before the administration of first dose of study intervention and must agree to use a highly-effective method of birth control.
* Participant is a non smoker or an ex-smoker with a total smoking history of less than 10 pack-years.
* Only for Part 1: Documented treatment with medium dose ICS with LABA for at least 6 months prior to Screening. ICS and LABA must be on a stable dose for at least 3 months prior to Screening, during Screening and Run-in Periods and may be contained in a combination product or separate inhaler. No asthma exacerbations in last 12 months requiring oral or intravenous (IV) steroids or hospitalisation/ emergency room visit due to asthma. Pre-bronchodilator FEV1 ≥ 70% predicted at Screening and start of Run-in. Asthma Control Questionnaire 6 score of ≤ 1.0 at Screening and start of Run-in.
* Only for Part 2: Documented evidence of asthma. Documented treatment with medium-to-high dose ICS-LABA for at least 6 months prior to Screening. ICS and LABA must be on a stable dose for at least 4 weeks prior to Screening, during Screening and Run-in Periods. If on asthma maintenance controller medications in addition to ICS-LABA, the dose of the additional controller medications must be stable for at least 4 weeks prior to Screening, during Screening and Run-in Periods. Pre bronchodilator FEV1 of 40% to 85% (inclusive) predicted at Screening and start of Run-in. Blood eosinophil count of ≥ 150 cells/μL and FeNO ≥ 25 ppb at Screening. Asthma Control Questionnaire 6 score ≥ 1.5 at Screening.

Specific Randomisation Criteria at Visit 3

* For Part 1: Pre-bronchodilator FEV1 ≥ 70% predicted. At least 70% compliance with usual asthma controller ICS-LABA during Run-in Period (from Visit 2 to Visit 3) based on daily electronic diary (e-Diary). Minimum 80% compliance with ePRO completion. Asthma Control Questionnaire 6 score of ≤ 1.0. C-reactive protein < 5 mg/L on Day -1.
* For Part 2: Pre-bronchodilator FEV1 of 40% to 85% (inclusive) predicted. Asthma Control Questionnaire 6 score of ≥ 1.5. At least 70% compliance with usual asthma controller ICS-LABA during Run-in Period from (Visit 2 to Visit 3) based on daily e-Diary. Minimum 70% compliance with ePRO completion. C-reactive protein < 10 mg/L at Visit 2. A FeNO of ≥ 25 ppb.

Exclusion Criteria:

* Women who are pregnant or breastfeeding, or who are planning to become pregnant during the study.
* Known or suspected hypersensitivity including anaphylaxis/anaphylactoid reaction following any biologic therapy, or known history of drug hypersensitivity to any component of the study intervention formulation.
* Evidence of any active clinically important pulmonary disease other than asthma, within 5 years at screening.
* History of pulmonary or systemic disease, other than asthma, that are associated with elevated peripheral eosinophil counts.
* History or clinical suspicion of any clinically relevant or active disease or disorder.
* History of severe COVID-19 infection requiring hospitalisation within the last 12 months or clinical history compatible with long COVID (symptoms beyond 12 weeks of acute infection).
* Confirmed symptomatic COVID-19 infection during Screening, Run-in or prior to randomisation.
* Current malignancy or history of malignancy.
* Significant history of recurrent or ongoing 'dry eye'.
* Diagnosis of Sjögren's syndrome.
* High risk of infection suggesting abnormal immune function.
* History of, or known significant infection or positivity at Screening period, including hepatitis B or C, or human immunodeficiency virus (HIV).
* Evidence of active tuberculosis.
* Clinically significant lower respiratory tract infection not resolved within 4 weeks prior to Screening and during Run-in.
* Clinically significant upper respiratory tract infection at Screening and during Run-in.
* A helminth parasitic infection diagnosed within 24 weeks prior to the date informed consent is obtained.
* Any clinically important ECG abnormalities.
* Any clinically significant cardiac disease.
* Uncontrolled hypertension.
* History of life-threatening asthma attack or asthma attack requiring ventilation.
* Part 2 only: History of 3 or more severe asthma exacerbations.
* Daily rescue use of SABA ≥ 8 puffs for ≥ 3 consecutive days at any time during Run-in Period, before randomisation.
* History of anaphylaxis.
* Any clinically significant abnormalities in haematology.
* Alanine aminotransferase or AST level ≥ 3 times the upper limit of normal (ULN), confirmed by repeated testing during Screening Period.
* History of, drug or alcohol abuse within the past 2 years prior to Screening.
* Planned in-patient surgery, major dental procedure or hospitalisation during the study.
* Prior/Concomitant Therapy: Systemic corticosteroid use, AZD1402, marketed or investigational biologicals such as monoclonal antibodies or chimeric biomolecules, investigational nonbiologic drug within 60 days prior to Screening and during Run-in, any immunosuppressive therapy, Live or attenuated vaccine within 4 weeks of Screening and during Run-in, Receipt of COVID-19 vaccine (vaccine or booster dose) within 30 days prior to randomisation, Immunoglobulin or blood products within 4 weeks of Screening and during Run-in, Any immunotherapy within 3 months of Screening and during Run-in.
* Part 1 only: Additional asthma maintenance controller medications in addition to ICS-LABA (eg, leukotriene receptor inhibitors, theophylline, LAMA, chromones) within 3 months of Screening period and during Run-in.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2021-03-12 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-07-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (32):
- Australia (3):
  - Research Site, Herston
  - Research Site, Melbourne
  - Research Site, Nedlands
- Canada (2):
  - Research Site, Windsor, Ontario
  - Research Site, Québec, Quebec
- Germany (6):
  - Research Site, Berlin
  - Research Site, Bonn
  - Research Site, Frankfurt
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Lübeck
- Hungary (2):
  - Research Site, Csorna
  - Research Site, Szombathely
- Poland (6):
  - Research Site, Bialystok
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Lubin
  - Research Site, Sopot
  - Research Site, Wroclaw
- South Korea (5):
  - Research Site, Cheongiu
  - Research Site, Incheon
  - Research Site, Namdong-gu
  - Research Site, Seoul
  - Research Site, Suwon
- Spain (3):
  - Research Site, Barcelona
  - Research Site, Santiago de Compostela
  - Research Site, Villarreal
- Research Site, Kaohsiung City, Taiwan
- Research Site, Kiev, Ukraine
- United Kingdom (3):
  - Research Site, High Wycombe
  - Research Site, Liverpool
  - Research Site, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in a sponsor approved tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D2912C00003&attachmentIdentifier=f7de1706-95c1-445e-b435-eec8003d0b38&fileName=D2912C00003-CSR_-Synopsis_1.0_dated_04Mar2024_Redacted.pdf&versionIdentifier=
- See also: CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D2912C00003&attachmentIdentifier=9d4ef8c9-6abc-43c1-8cac-fdf4dacf6ef7&fileName=d2912c00003-csp-v8-signed_Redacted.pdf&versionIdentifier=
- See also: SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D2912C00003&attachmentIdentifier=47315e15-4c7f-45c9-914d-f8f206665ff4&fileName=d2912c00003-sap-ed-5_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted from 21 April 2021 to 20 July 2023 at 63 study centers in 10 countries.
Pre-assignment Details: The screening period was of 2 weeks (Week -6 to Week -4) for both parts of the study. Informed Consent Form (ICF) was signed prior to screening procedures. All the study assessments were performed as per the schedule of assessment. Participants who met the eligibility criteria were randomized to study intervention in addition to receiving background local standard of care therapy.
Groups:
- Part 1: AZD1402 Dose 1: Randomised participants received oral inhalation of AZD1402 Dose 1 via dry powder inhaler (DPI).
- Part 1: AZD1402 Dose 2; Part 2: AZD1402 Dose 2: Randomised participants received oral inhalation of AZD1402 Dose 2 via DPI.
- Part 1: AZD1402 Dose 3: Randomised participants received oral inhalation of AZD1402 Dose 3 via DPI.
- Part 1: Placebo; Part 2: Placebo: Randomised participants received oral inhalation of matching placebo via DPI.
- Part 2: AZD1402 Dose 1: Randomised participants received oral inhalation of AZD1402 Dose 1 via DPI.
Period: Overall Study
Arm/Group | Part 1: AZD1402 Dose 1 | Part 1: AZD1402 Dose 2 | Part 1: AZD1402 Dose 3 | Part 1: Placebo | Part 2: AZD1402 Dose 1 | Part 2: AZD1402 Dose 2 | Part 2: Placebo
Started | 11 | 10 | 13 | 16 | 4 | 9 | 9
Completed | 11 | 10 | 11 | 16 | 4 | 7 | 9
Not Completed | 0 | 0 | 2 | 0 | 0 | 2 | 0
Not completed — Study terminated by sponsor | 0 | 0 | 1 | 0 | 0 | 1 | 0
Not completed — Global/country situation | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set included all patients who were randomised and received any investigational product (IP).
Groups:
- Part 1: AZD1402 Dose 1; Part 2: AZD1402 Dose 1: Randomised participants received oral inhalation of AZD1402 Dose 1 via DPI.
- Total: Total of all reporting groups
Arm/Group | Part 1: AZD1402 Dose 1 | Part 1: AZD1402 Dose 2 | Part 1: AZD1402 Dose 3 | Part 1: Placebo | Part 2: AZD1402 Dose 1 | Part 2: AZD1402 Dose 2 | Part 2: Placebo | Total
Number analyzed (Participants) | 11 | 10 | 13 | 16 | 4 | 9 | 9 | 72
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.3 (11.5) | 43.6 (15.2) | 47.0 (17.6) | 50.0 (10.8) | 60.3 (10.2) | 61.3 (6.5) | 61.7 (6.6) | 52.9 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 7 | 8 | 2 | 6 | 4 | 40
  Male | 4 | 4 | 6 | 8 | 2 | 3 | 5 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 11 | 10 | 13 | 16 | 4 | 8 | 9 | 71
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants With Adverse Events (AEs)
Description: The safety and tolerability of AZD1402 compared to placebo at different dose levels in adults with asthma controlled on medium dose ICS-LABA was evaluated.
Time Frame: From Screening (Week -6) until Follow-up (Day 56)
Population: The safety set included all patients who were randomised and received any investigational product (IP).
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: AZD1402 Dose 1 | Part 1: AZD1402 Dose 2 | Part 1: AZD1402 Dose 3 | Part 1: Placebo
Number analyzed (Participants) | 11 | 10 | 13 | 16
Participants
  Any AE | 4 | 6 | 10 | 8
  Any SAE | 0 | 0 | 0 | 0
  Any SAE with outcome death | 0 | 0 | 0 | 0
  Any AE leading to discontinuation of IP | 0 | 1 | 1 | 1
  Any AE leading to withdrawal from study | 0 | 0 | 0 | 0

2. Primary Outcome: Part 2: Change From Baseline in Pre-bronchodilator FEV1
Description: The efficacy of inhaled AZD1402 compared to placebo in adults with asthma uncontrolled on medium-to-high dose ICS-LABA was investigated.
Time Frame: Baseline and Week 4
Population: The full analysis set included all patients who were randomised and received any IP.
Measure: Least Squares Mean (Standard Error); unit: Liters (L)
Arm/Group | Part 2: AZD1402 Dose 1 | Part 2: AZD1402 Dose 2 | Part 2: Placebo
Number analyzed (Participants) | 4 | 9 | 9
Liters (L) | -0.0195 (0.1023) | 0.1529 (0.0804) | -0.0431 (0.0777)
Statistical Analysis 1: Comparison: Part 2: AZD1402 Dose 1 vs Part 2: Placebo; Test type: Superiority; p = 0.828, Mixed Models Analysis; Least Square Mean Difference = 0.0236, 95% CI 2-sided [-0.1934 to 0.2406]
Statistical Analysis 2: Comparison: Part 2: AZD1402 Dose 2 vs Part 2: Placebo; Test type: Superiority; p = 0.035, Mixed Models Analysis; Least Square Mean Difference = 0.1960, 95% CI 2-sided [0.0143 to 0.3778]

3. Secondary Outcome: Part 1 and Part 2: Antidrug Antibodies (ADA) Titers
Description: ADA-positive samples were tested to investigate the immunogenicity of AZD1402.
Time Frame: Day 1 until Day 56
Population: The immunogenicity set included all participants in the safety set with at least one post-treatment ADA result (positive or negative). Here, 'number of participants analyzed' specifies participants evaluated for this outcome measure at specific timepoints. Participants in the Part 1: Placebo arm did not have any post-treatment ADA results and were excluded from analysis.
Measure: Median (Inter-Quartile Range); unit: Titer
Arm/Group | Part 1: AZD1402 Dose 1 | Part 1: AZD1402 Dose 2 | Part 1: AZD1402 Dose 3 | Part 1: Placebo | Part 2: AZD1402 Dose 1 | Part 2: AZD1402 Dose 2 | Part 2: Placebo
Number analyzed (Participants) | 10 | 10 | 8 | 0 | 4 | 6 | 6
Titer
  ADA positive at baseline and/or post-baseline (ADA prevalence): number analyzed (Participants) | 10 | 10 | 8 | 0 | 4 | 6 | 0
  ADA positive at baseline and/or post-baseline (ADA prevalence) | 1280.0 [160.0 to 5120.0] | 360.0 [40.0 to 1280.0] | 320.0 [240.0 to 800.0] |  | 240.0 [90.0 to 800.0] | 400.0 [160.0 to 2560.0] |
  TE-ADA positive (ADA incidence): number analyzed (Participants) | 10 | 10 | 8 | 0 | 4 | 6 | 0
  TE-ADA positive (ADA incidence) | 1280.0 [160.0 to 5120.0] | 360.0 [40.0 to 1280.0] | 320.0 [240.0 to 800.0] |  | 240.0 [90.0 to 800.0] | 400 [160.0 to 2560.0] |
  Treatment-induced ADA positive: number analyzed (Participants) | 10 | 10 | 8 | 0 | 4 | 6 | 0
  Treatment-induced ADA positive | 1280.0 [160.0 to 5120.0] | 360.0 [40.0 to 1280.0] | 320.0 [240.0 to 800.0] |  | 240.0 [90.0 to 800.0] | 400 [160.0 to 2560.0] |
  ADA persistently positive: number analyzed (Participants) | 10 | 9 | 8 | 0 | 0 | 4 | 6
  ADA persistently positive | 1280.0 [160.0 to 5120.0] | 640.0 [80.0 to 1280.0] | 320.0 [240.0 to 800.0] |  |  | 240.0 [90.0 to 800.0] | 400.0 [160.0 to 2560.0]
  ADA transiently positive: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0
  ADA transiently positive |  | NA [NA to NA] — Values are not calculated due to insufficient number of participants with events. |  |  |  |  |
  TE-ADA positive with maximum titre > median of maximum titres: number analyzed (Participants) | 6 | 5 | 2 | 0 | 1 | 3 | 0
  TE-ADA positive with maximum titre > median of maximum titres | 3840.0 [1280.0 to 5120.0] | 1280.0 [640.0 to 1280.0] | NA [NA to NA] — Values are not calculated due to insufficient number of participants with events. |  | NA — Values are not calculated due to insufficient number of participants with events. | 2560.0 [640.0 to 2560.9] |

4. Secondary Outcome: Part 1 and Part 2: Maximum Observed Serum (Peak) Drug Concentration (Cmax)
Description: The pharmacokinetic (PK) profile of AZD1402 was investigated.
Time Frame: Day 1 until Day 56
Population: The PK set included all patients in the safety set who had detectable PK data and with no major protocol deviations considered to impact on the analysis of PK data. Here, 'number of participants analyzed' specifies participants evaluated for this outcome measure at specific timepoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms Per Milliliter (ng/mL)
Arm/Group | Part 1: AZD1402 Dose 1 | Part 1: AZD1402 Dose 2 | Part 1: AZD1402 Dose 3 | Part 2: AZD1402 Dose 1 | Part 2: AZD1402 Dose 2
Number analyzed (Participants) | 8 | 8 | 11 | 4 | 7
Nanograms Per Milliliter (ng/mL)
  Day 1: number analyzed (Participants) | 2 | 8 | 11 | 4 | 7
  Day 1 | NA (NA) — Values are not calculated due to insufficient number of participants with data. | 2.745 (43.2) | 5.864 (50.2) | NA (NA) — Values below the lower limit of quantification are not calculated. | NA (NA) — Values below the lower limit of quantification are not calculated.
  Day 28: number analyzed (Participants) | 8 | 8 | 10 | 4 | 7
  Day 28 | 3.986 (68.9) | 10.46 (103.0) | 30.97 (124.7) | NA (NA) — Values below the lower limit of quantification are not calculated. | NA (NA) — Values below the lower limit of quantification are not calculated.

5. Secondary Outcome: Part 1 and Part 2: Half-life Associated With Terminal Slope (λz) of a Semi-logarithmic Concentration-time Curve (t1/2λz)
Description: The PK profile of AZD1402 was investigated.
Time Frame: Day 1 until Day 56
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours (h)
Arm/Group | Part 1: AZD1402 Dose 1 | Part 1: AZD1402 Dose 2 | Part 1: AZD1402 Dose 3 | Part 2: AZD1402 Dose 1 | Part 2: AZD1402 Dose 2
Number analyzed (Participants) | 6 | 7 | 10 | 4 | 7
Hours (h)
  Day 1: number analyzed (Participants) | 0 | 2 | 7 | 4 | 7
  Day 1 |  | NA (NA) — Values are not calculated due to insufficient number of participants with data. | 9.440 (49.4) | NA (NA) — Values below the lower limit of quantification are not calculated. | NA (NA) — Values below the lower limit of quantification are not calculated.
  Day 28 | 20.17 (668.7) | 7.669 (33.2) | 8.546 (34.5) | NA (NA) — Values below the lower limit of quantification are not calculated. | NA (NA) — Values below the lower limit of quantification are not calculated.

6. Secondary Outcome: Part 1 and Part 2: Area Under Plasma Concentration-time Curve in the Dosing Interval τ (AUCτ)
Description: The PK profile of AZD1402 was investigated.
Time Frame: Day 1 until Day 56
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part 1: AZD1402 Dose 1 | Part 1: AZD1402 Dose 2 | Part 1: AZD1402 Dose 3 | Part 2: AZD1402 Dose 1 | Part 2: AZD1402 Dose 2
Number analyzed (Participants) | 8 | 8 | 11 | 4 | 7
h*ng/mL
  Day 1: number analyzed (Participants) | 0 | 4 | 11 | 4 | 7
  Day 1 |  | 23.15 (28.9) | 46.34 (52.4) | NA (NA) — Values below the lower limit of quantification are not calculated. | NA (NA) — Values below the lower limit of quantification are not calculated.
  Day 28: number analyzed (Participants) | 6 | 8 | 10 | 4 | 7
  Day 28 | 46.75 (63.3) | 92.80 (94.4) | 264.4 (132.7) | NA (NA) — Values below the lower limit of quantification are not calculated. | NA (NA) — Values below the lower limit of quantification are not calculated.

7. Secondary Outcome: Part 1 and Part 2: Area Under the Plasma Concentration-curve From Zero to the Last Quantifiable Concentration (AUClast)
Description: The PK profile of AZD1402 was investigated.
Time Frame: Day 1 until Day 56
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part 1: AZD1402 Dose 1 | Part 1: AZD1402 Dose 2 | Part 1: AZD1402 Dose 3 | Part 2: AZD1402 Dose 1 | Part 2: AZD1402 Dose 2
Number analyzed (Participants) | 8 | 8 | 11 | 4 | 7
h*ng/mL
  Day 1: number analyzed (Participants) | 0 | 6 | 11 | 4 | 7
  Day 1 |  | 16.32 (57.8) | 44.40 (56.9) | NA (NA) — Values below the lower limit of quantification are not calculated. | NA (NA) — Values below the lower limit of quantification are not calculated.
  Day 28: number analyzed (Participants) | 8 | 8 | 10 | 4 | 7
  Day 28 | 44.26 (604.9) | 146.3 (144.7) | 379.4 (169.6) | NA (NA) — Values below the lower limit of quantification are not calculated. | NA (NA) — Values below the lower limit of quantification are not calculated.

8. Secondary Outcome: Part 1 and Part 2: Observed Lowest Drug Concentration Reached Before the Next Dose is Administered (Pre-dose) (Ctrough)
Description: The PK profile of AZD1402 was investigated.
Time Frame: Day 1 until Day 56
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1: AZD1402 Dose 1 | Part 1: AZD1402 Dose 2 | Part 1: AZD1402 Dose 3 | Part 2: AZD1402 Dose 1 | Part 2: AZD1402 Dose 2
Number analyzed (Participants) | 6 | 8 | 10 | 4 | 7
ng/mL
  Day 1: number analyzed (Participants) | 0 | 4 | 7 | 4 | 7
  Day 1 |  | 1.702 (30.0) | 2.917 (53.6) | NA (NA) — Values below the lower limit of quantification are not calculated. | NA (NA) — Values below the lower limit of quantification are not calculated.
  Day 28 | 2.854 (66.3) | 5.145 (96.8) | 13.83 (144.2) | NA (NA) — Values below the lower limit of quantification are not calculated. | NA (NA) — Values below the lower limit of quantification are not calculated.

9. Secondary Outcome: Part 1 and Part 2: Terminal Rate Constant, Estimated by Log-linear Least Squares Regression of the Terminal Part of the Concentration-time Curve (λz)
Description: The PK profile of AZD1402 was investigated.
Time Frame: Day 1 until Day 56
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hour
Arm/Group | Part 1: AZD1402 Dose 1 | Part 1: AZD1402 Dose 2 | Part 1: AZD1402 Dose 3 | Part 2: AZD1402 Dose 1 | Part 2: AZD1402 Dose 2
Number analyzed (Participants) | 6 | 7 | 10 | 4 | 7
1/hour
  Day 1: number analyzed (Participants) | 0 | 2 | 7 | 4 | 7
  Day 1 |  | NA (NA) — Values are not calculated due to insufficient number of participants with data. | 0.07343 (49.4) | NA (NA) — Values below the lower limit of quantification are not calculated. | NA (NA) — Values below the lower limit of quantification are not calculated.
  Day 28 | 0.03437 (668.7) | 0.09040 (33.2) | 0.08111 (34.5) | NA (NA) — Values below the lower limit of quantification are not calculated. | NA (NA) — Values below the lower limit of quantification are not calculated.

10. Secondary Outcome: Part 1 and Part 2: Volume of Distribution (Apparent) at Steady State Following Extravascular Administration (Based on Terminal Phase) (Vz/F)
Description: The PK profile of AZD1402 was investigated.
Time Frame: Day 1 until Day 56
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Part 1: AZD1402 Dose 1 | Part 1: AZD1402 Dose 2 | Part 1: AZD1402 Dose 3 | Part 2: AZD1402 Dose 1 | Part 2: AZD1402 Dose 2
Number analyzed (Participants) | 6 | 7 | 10 | 4 | 7
Liters | 622.5 (1007.5) | 322.9 (109.7) | 466.3 (172.0) | NA (NA) — Values below the lower limit of quantification are not calculated. | NA (NA) — Values below the lower limit of quantification are not calculated.

11. Secondary Outcome: Part 1 and Part 2: Apparent Total Body Clearance of Drug From Plasma After Extravascular Administration (CL/F)
Description: The PK profile of AZD1402 was investigated.
Time Frame: Day 1 until Day 56
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters/hour (L/h)
Arm/Group | Part 1: AZD1402 Dose 1 | Part 1: AZD1402 Dose 2 | Part 1: AZD1402 Dose 3 | Part 2: AZD1402 Dose 1 | Part 2: AZD1402 Dose 2
Number analyzed (Participants) | 6 | 8 | 10 | 4 | 7
Liters/hour (L/h) | 21.39 (63.3) | 32.33 (94.4) | 37.82 (132.7) | NA (NA) — Values below the lower limit of quantification are not calculated. | NA (NA) — Values below the lower limit of quantification are not calculated.

12. Secondary Outcome: Part 1 and Part 2: Time to Reach Peak or Maximum Observed Concentration or Response Following Drug Administration (Tmax)
Description: The PK profile of AZD1402 was investigated.
Time Frame: Day 1 until Day 56
Population: as for outcome 4
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: AZD1402 Dose 1 | Part 1: AZD1402 Dose 2 | Part 1: AZD1402 Dose 3 | Part 2: AZD1402 Dose 1 | Part 2: AZD1402 Dose 2
Number analyzed (Participants) | 8 | 8 | 11 | 1 | 2
Hours
  Day 1: number analyzed (Participants) | 2 | 8 | 11 | 0 | 1
  Day 1 | NA [3.00 to 6.00] — Values are not calculated due to insufficient number of participants with data. | 3.000 [2.00 to 8.00] | 4.017 [3.02 to 8.02] |  | NA [3.05 to 3.05] — Values are not calculated due to insufficient number of participants with data.
  Day 28: number analyzed (Participants) | 8 | 8 | 10 | 1 | 2
  Day 28 | 3.025 [1.00 to 4.00] | 3.000 [0.00 to 6.00] | 3.950 [3.00 to 6.27] | NA [5.93 to 5.93] — Values are not calculated due to insufficient number of participants with data. | NA [7.67 to 8.07] — Values are not calculated due to insufficient number of participants with data.

13. Secondary Outcome: Part 1 and Part 2: Time of Last Observed (Quantifiable) Concentration (Tlast)
Description: The PK profile of AZD1402 was investigated.
Time Frame: Day 1 until Day 56
Population: as for outcome 4
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: AZD1402 Dose 1 | Part 1: AZD1402 Dose 2 | Part 1: AZD1402 Dose 3 | Part 2: AZD1402 Dose 1 | Part 2: AZD1402 Dose 2
Number analyzed (Participants) | 8 | 8 | 11 | 1 | 2
Hours
  Day 1: number analyzed (Participants) | 2 | 8 | 11 | 0 | 1
  Day 1 | NA [3.00 to 8.00] — Values are not calculated due to insufficient number of participants with data. | 8.000 [2.00 to 12.0] | 11.47 [8.18 to 12.0] |  | NA [6.97 to 6.97] — Values are not calculated due to insufficient number of participants with data.
  Day 28: number analyzed (Participants) | 8 | 8 | 10 | 1 | 2
  Day 28 | 11.99 [3.00 to 576] | 17.83 [12.0 to 48.2] | 23.94 [12.0 to 47.9] | NA [5.93 to 5.93] — Values are not calculated due to insufficient number of participants with data. | NA [7.67 to 22.8] — Values are not calculated due to insufficient number of participants with data.

14. Secondary Outcome: Part 1 and Part 2: Accumulation Ratio for AUCτ (Rac AUC)
Description: The PK profile of AZD1402 was investigated.
Time Frame: Day 1 until Day 56
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Part 1: AZD1402 Dose 1 | Part 1: AZD1402 Dose 2 | Part 1: AZD1402 Dose 3 | Part 2: AZD1402 Dose 1 | Part 2: AZD1402 Dose 2
Number analyzed (Participants) | 1 | 3 | 8 | 4 | 7
Ratio | NA (NA) — Values below the lower limit of quantification are not calculated. | NA (NA) — Values are not calculated due to insufficient number of participants with data. | 6.059 (68.5) | NA (NA) — Values below the lower limit of quantification are not calculated. | NA (NA) — Values below the lower limit of quantification are not calculated.

15. Secondary Outcome: Part 1 and Part 2: Accumulation Ratio for Cmax (Rac Cmax)
Description: The PK profile of AZD1402 was investigated.
Time Frame: Day 1 until Day 56
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Part 1: AZD1402 Dose 1 | Part 1: AZD1402 Dose 2 | Part 1: AZD1402 Dose 3 | Part 2: AZD1402 Dose 1 | Part 2: AZD1402 Dose 2
Number analyzed (Participants) | 2 | 6 | 8 | 4 | 7
Ratio | NA (NA) — Values are not calculated due to insufficient number of participants with data. | 3.219 (121.9) | 6.067 (78.9) | NA (NA) — Values below the lower limit of quantification are not calculated. | NA (NA) — Values below the lower limit of quantification are not calculated.

16. Secondary Outcome: Part 2: Change From Baseline in Asthma Control Questionnaire-6 (ACQ-6) at Week 4 and Average Over the Treatment Period
Description: The efficacy of AZD1402 compared to placebo in adults with asthma who are uncontrolled on medium-to-high dose ICS-LABA was further investigated. The ACQ was developed to measure asthma control. In the ACQ-6, participants were asked to recall how their asthma had been during the previous week by responding to one bronchodilation use question and 5 symptom questions. Questions were weighted equally and scored from 0 (totally controlled) to 6 (severely uncontrolled). Higher scores indicated a worse outcome. The mean ACQ-6 score is the mean of the responses. Mean scores of ≤ 0.75 indicate well-controlled asthma, scores between 0.75 and ≤ 1.5 indicate partly controlled asthma, and scores > 1.5 indicate not well-controlled asthma. Individual changes of at least 0.5 are considered clinically meaningful.
Time Frame: Baseline, Week 4
Population: The full analysis set included all patients who were randomised and received any IP. Here, 'number of participants analyzed' specifies participants evaluated for this outcome measure at specific timepoints.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Part 2: AZD1402 Dose 1 | Part 2: AZD1402 Dose 2 | Part 2: Placebo
Number analyzed (Participants) | 4 | 9 | 9
Score on scale
  Change from baseline at Week 4 | -0.80 (0.37) | -0.71 (0.68) | -0.56 (0.75)
  Average change from baseline over treatment period | -0.75 (0.56) | -0.78 (0.33) | -0.56 (0.66)

17. Secondary Outcome: Part 2: Participants With a Decrease in ACQ 6 Score of ≥ 0.5 From Baseline to Week 4
Description: as for outcome 16
Time Frame: Baseline, Week 4
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: AZD1402 Dose 1 | Part 2: AZD1402 Dose 2 | Part 2: Placebo
Number analyzed (Participants) | 4 | 9 | 9
Participants
  Responder | 3 | 7 | 3
  Non-responder | 1 | 2 | 6

18. Secondary Outcome: Part 2: Change From Baseline in Average Morning Peak Expiratory Flow (PEF) Over the Treatment Period
Description: The efficacy of AZD1402 compared to placebo in adults with asthma uncontrolled on medium-to-high dose ICS-LABA was further investigated. Peak expiratory flow was measured by the participants at home using a peak flow meter.
Time Frame: Baseline, 4 weeks
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Liters/minute (L/m)
Arm/Group | Part 2: AZD1402 Dose 1 | Part 2: AZD1402 Dose 2 | Part 2: Placebo
Number analyzed (Participants) | 4 | 9 | 9
Liters/minute (L/m)
  Change from baseline at Week 4 | 23.73 (15.24) | 19.88 (47.38) | -2.53 (26.69)
  Average change from baseline over the treatment period | 20.67 (8.58) | 21.40 (37.83) | -5.54 (24.17)

19. Secondary Outcome: Part 2: Change From Baseline in Average Evening PEF Over the Treatment Period
Description: as for outcome 18
Time Frame: Baseline, 4 weeks
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Liters/minute (L/m)
Arm/Group | Part 2: AZD1402 Dose 1 | Part 2: AZD1402 Dose 2 | Part 2: Placebo
Number analyzed (Participants) | 4 | 9 | 9
Liters/minute (L/m)
  Change from baseline at Week 4 | 18.68 (3.94) | -15.81 (28.63) | 0.89 (30.22)
  Average change from baseline over the treatment period | 14.20 (10.37) | -7.75 (25.79) | 1.87 (19.27)

20. Secondary Outcome: Part 2: Change From Baseline in Daily Average Asthma Symptom Score (AM/PM) Over the Treatment Period
Description: The efficacy of AZD1402 compared to placebo in adults with asthma uncontrolled on medium-to-high dose ICS-LABA was further investigated. Severity scores for asthma symptoms were recorded twice daily in the morning and evening and documented in an e-Diary. Asthma symptom scores during night-time and day-time were assessed by the participant each morning and evening according to the following scoring system: 0: You have no asthma symptoms. 1: You are aware of your asthma symptoms but you can easily tolerate the symptoms. 2: Your asthma is causing you enough discomfort to cause problems with normal activities (or with sleep). 3: You are unable to do your normal activities (or to sleep) because of your asthma. Higher scores indicated worse outcome.
Time Frame: Baseline, 4 weeks
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Part 2: AZD1402 Dose 1 | Part 2: AZD1402 Dose 2 | Part 2: Placebo
Number analyzed (Participants) | 4 | 9 | 9
Score on scale
  Change from baseline at Week 4 | -0.23 (0.26) | 0.07 (0.26) | -0.04 (0.37)
  Average change from baseline over the treatment period | -0.10 (0.27) | 0.02 (0.22) | -0.07 (0.32)

21. Secondary Outcome: Part 2: Change From Baseline in Pre-bronchodilator FEV1 Average Over the 4-week Treatment Period
Description: The efficacy of AZD1402 compared to placebo in adults with asthma uncontrolled on medium-to-high dose ICS-LABA was further investigated.
Time Frame: Baseline and Week 4
Population: as for outcome 16
Measure: Least Squares Mean (Standard Error); unit: Liters (L)
Arm/Group | Part 2: AZD1402 Dose 1 | Part 2: AZD1402 Dose 2 | Part 2: Placebo
Number analyzed (Participants) | 4 | 9 | 9
Liters (L)
  Week 1: number analyzed (Participants) | 4 | 9 | 8
  Week 1 | 0.0233 (0.0526) | 0.1408 (0.1679) | 0.0101 (0.1094)
  Week 2: number analyzed (Participants) | 4 | 8 | 9
  Week 2 | 0.0028 (0.0618) | 0.0866 (0.1607) | 0.1671 (0.3323)
  Week 3 | 0.0160 (0.1140) | 0.0431 (0.1676) | 0.1099 (0.1583)
  Week 4 | 0.0095 (0.1085) | 0.1500 (0.1898) | -0.0252 (0.1754)

22. Secondary Outcome: Part 2: Change From Baseline in FeNO (In-clinic) at Week 4 and Average Over the Treatment Period
Description: The effect of AZD1402 compared to placebo on airway inflammation in adults with asthma uncontrolled on medium-to-high dose ICS-LABA was investigated. To investigate the effect of AZD1402 on airway inflammation, the measurement of FeNO was performed in accordance with ATS/ERS guidelines. Standardised conditions with regard to exhalation flow rate and duration of exhalation were followed such that plateau definition could be evaluated over a minimum of 3 seconds.
Time Frame: Baseline, Week 4
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Parts per billion (ppb)
Arm/Group | Part 2: AZD1402 Dose 1 | Part 2: AZD1402 Dose 2 | Part 2: Placebo
Number analyzed (Participants) | 4 | 9 | 9
Parts per billion (ppb)
  Change from baseline at Week 4 | 39.77 (55.03) | 28.76 (91.99) | 31.20 (122.50)
  Average change from baseline over the treatment period | 32.02 (153.61) | 14.16 (343.96) | 27.45 (102.83)
Statistical Analysis 1: Comparison: Part 2: AZD1402 Dose 1 vs Part 2: Placebo; Test type: Superiority; p = 0.202, Mixed Models Analysis; Geometric Least Square Mean Ratio = -38.31, 95% CI 2-sided [-71.11 to 31.72] — Analyses were done on the natural log scale and the results were back-transformed to linear scale
Statistical Analysis 2: Comparison: Part 2: AZD1402 Dose 2 vs Part 2: Placebo; Test type: Superiority; p = 0.596, Mixed Models Analysis; Geometric Least Square Mean Ratio = -15.43, 95% CI 2-sided [-55.57 to 60.96] — Analyses were done on the natural log scale and the results were back-transformed to linear scale

23. Secondary Outcome: Part 2: Number of Participants With Adverse Events (AEs)
Description: The safety and tolerability of AZD1402 compared to placebo in adults with asthma uncontrolled on medium-to-high dose ICS-LABA was evaluated.
Time Frame: From Screening (Week -6) until Follow-up (Day 56)
Population: The safety set included all patients who were randomised and received any IP. Here, 'number of participants analyzed' specifies participants evaluated for this outcome measure at specific timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: AZD1402 Dose 1 | Part 2: AZD1402 Dose 2 | Part 2: Placebo
Number analyzed (Participants) | 4 | 9 | 9
Participants
  Any AE | 3 | 5 | 6
  Any SAE | 0 | 1 | 0
  Any SAE with outcome death | 0 | 0 | 0
  Any AE leading to discontinuation of IP | 0 | 0 | 0
  Any AE leading to withdrawal from study | 0 | 0 | 0

24. Primary Outcome: Part 1: Change From Baseline in High-sensitivity C-reactive Protein (hsCRP)
Description: as for outcome 1
Time Frame: Baseline, Day 12, Day 16, and Day 56
Population: The safety set included all patients who were randomised and received any IP.
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | Part 1: AZD1402 Dose 1 | Part 1: AZD1402 Dose 2 | Part 1: AZD1402 Dose 3 | Part 1: Placebo
Number analyzed (Participants) | 11 | 10 | 13 | 16
milligrams per deciliter (mg/dL)
  Baseline | 0.225 (0.369) | 0.109 (0.080) | 0.102 (0.070) | 0.094 (0.090)
  Day 12: number analyzed (Participants) | 11 | 10 | 12 | 16
  Day 12 | 0.167 (0.247) | 0.650 (1.898) | 0.485 (0.542) | 0.103 (0.173)
  Day 16: number analyzed (Participants) | 11 | 9 | 12 | 16
  Day 16 | 0.727 (1.906) | 0.166 (0.171) | 1.093 (1.761) | 0.088 (0.091)
  Day 56: number analyzed (Participants) | 11 | 10 | 11 | 15
  Day 56 | 0.172 (0.243) | 0.094 (0.095) | 0.119 (0.081) | 0.112 (0.151)

25. Primary Outcome: Part 1: Change From Baseline in FEV1 In-clinic Spirometry
Description: as for outcome 1
Time Frame: Baseline, Day 1, Day 7, Day 14, Day 28, and Day 56
Population: The safety set included all patients who were randomised and received any IP.
Measure: Mean (Standard Deviation); unit: Liters (L)
Arm/Group | Part 1: AZD1402 Dose 1 | Part 1: AZD1402 Dose 2 | Part 1: AZD1402 Dose 3 | Part 1: Placebo
Number analyzed (Participants) | 11 | 10 | 13 | 16
Liters (L)
  Day 1 evening: number analyzed (Participants) | 11 | 10 | 12 | 16
  Day 1 evening | -0.0338 (0.1794) | -0.2416 (0.4113) | 0.0031 (0.1841) | 0.0318 (0.1362)
  Day 7 morning: number analyzed (Participants) | 11 | 10 | 12 | 16
  Day 7 morning | -0.1225 (0.1290) | -0.2134 (0.1975) | 0.0187 (0.1338) | -0.0913 (0.2121)
  Day 7 evening: number analyzed (Participants) | 11 | 10 | 12 | 16
  Day 7 evening | -0.0648 (0.1579) | -0.0884 (0.1082) | 0.0430 (0.1613) | 0.0486 (0.1474)
  Day 14 morning: number analyzed (Participants) | 11 | 10 | 12 | 16
  Day 14 morning | -0.1157 (0.1231) | -0.1776 (0.1533) | -0.0388 (0.2225) | -0.0773 (0.1584)
  Day 28 morning: number analyzed (Participants) | 10 | 9 | 11 | 14
  Day 28 morning | -0.2199 (0.1933) | -0.1673 (0.2192) | -0.0583 (0.1515) | -0.2050 (0.2290)
  Day 56: number analyzed (Participants) | 11 | 10 | 11 | 15
  Day 56 | -0.2239 (0.2096) | -0.1232 (0.1455) | -0.0830 (0.1802) | -0.1707 (0.2345)

26. Primary Outcome: Part 1: Change From Baseline in Fractional Exhaled Nitric Oxide (FeNO) (In-clinic)
Description: as for outcome 1
Time Frame: Baseline, Day 1, Day 7, Day 14, Day 28, and Day 56
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Part per billion (ppb)
Arm/Group | Part 1: AZD1402 Dose 1 | Part 1: AZD1402 Dose 2 | Part 1: AZD1402 Dose 3 | Part 1: Placebo
Number analyzed (Participants) | 11 | 10 | 13 | 16
Part per billion (ppb)
  Day 1 evening: number analyzed (Participants) | 11 | 10 | 12 | 16
  Day 1 evening | 12.14 (123.28) | 17.14 (356.42) | 13.52 (162.23) | 13.30 (150.60)
  Day 7 morning: number analyzed (Participants) | 11 | 10 | 12 | 16
  Day 7 morning | 11.60 (243.83) | 23.71 (132.90) | 21.55 (95.95) | 17.61 (93.96)
  Day 7 evening: number analyzed (Participants) | 11 | 10 | 12 | 16
  Day 7 evening | 16.81 (102.28) | 18.83 (230.59) | 22.97 (155.86) | 16.90 (140.49)
  Day 14 morning: number analyzed (Participants) | 11 | 10 | 12 | 16
  Day 14 morning | 18.17 (213.64) | 23.17 (204.29) | 25.06 (168.79) | 31.32 (183.61)
  Day 28 morning: number analyzed (Participants) | 10 | 9 | 11 | 14
  Day 28 morning | 19.07 (143.18) | 16.31 (170.18) | 20.06 (289.93) | 16.50 (148.92)
  Day 56 morning: number analyzed (Participants) | 11 | 10 | 11 | 15
  Day 56 morning | 14.17 (174.36) | 19.31 (62.10) | 21.44 (212.81) | 15.51 (106.64)
  Average change from baseline over the treatment period | 10.23 (164.24) | 16.37 (183.76) | 20.78 (111.33) | 14.60 (127.31)

ADVERSE EVENTS:
Time Frame: From Screening (Week -6) until Follow-up (Day 56)
Arm/Group | Part 1: AZD1402 Dose 1 | Part 1: AZD1402 Dose 2 | Part 1: AZD1402 Dose 3 | Part 1: Placebo | Part 2: AZD1402 Dose 1 | Part 2: AZD1402 Dose 2 | Part 2: Placebo
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/10 | 0/13 | 0/16 | 0/4 | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10 | 0/13 | 0/16 | 0/4 | 1/9 | 0/9
Other Adverse Events (participants affected / at risk) | 4/11 | 6/10 | 10/13 | 8/16 | 3/4 | 5/9 | 6/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: AZD1402 Dose 1 (N=11) | Part 1: AZD1402 Dose 2 (N=10) | Part 1: AZD1402 Dose 3 (N=13) | Part 1: Placebo (N=16) | Part 2: AZD1402 Dose 1 (N=4) | Part 2: AZD1402 Dose 2 (N=9) | Part 2: Placebo (N=9)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: AZD1402 Dose 1 (N=11) | Part 1: AZD1402 Dose 2 (N=10) | Part 1: AZD1402 Dose 3 (N=13) | Part 1: Placebo (N=16) | Part 2: AZD1402 Dose 1 (N=4) | Part 2: AZD1402 Dose 2 (N=9) | Part 2: Placebo (N=9)
Covid-19 (Infections and infestations) | 0 | 1 | 0 | 1 | 1 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1 | 3 | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 5 | 0 | 1 | 0 | 0
Tension headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Conjuctivitis allergic (Eye disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Ear haemorrhage (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 4 | 3 | 1 | 0 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 5 | 2 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 3 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3 | 0 | 0 | 0 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Leukocyturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
C-reactive protein increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Forced expiratory volume decreased (Investigations) | 2 | 3 | 1 | 1 | 0 | 0 | 0
Transaminases (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood thyroid stimulating hormone decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bone contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Terminated (The decision was based on lung findings from a non-clinical 13-week Good Laboratory Practice (GLP) toxicology study, which are not a concern for the active clinical studies but do not support long-term use and progression to later-stage development).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
This document contains trade secrets and confidential commercial information, disclosure of which is prohibited without providing advance notice to AstraZeneca and opportunity to object.

DOCUMENTS (2):
  • Study Protocol (2023-03-24): https://cdn.clinicaltrials.gov/large-docs/58/NCT04643158/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-26): https://cdn.clinicaltrials.gov/large-docs/58/NCT04643158/SAP_001.pdf